CLINICAL TRIAL: NCT05975112
Title: The Incidence of Hyperfibrinolysis During Vaginal Delivery and Cesarean Section
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 13
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Hyperfibrinolysis; Cesarean Section Complications; Coagulation Defect; Bleeding; Peripartum Haemorrhage
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — one blood sample of 6ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cesarean section: maternal blood is drawn immediately after the baby's cord is cut and analyzed using thrombelastography with the addition of tranexamic acid. In addition, the following parameters are examined:
  * Levels of Factor 1 (Fibrinogen) and Factor 2 (Thrombin)
  * Level of hs-D-Dimer
  SpHb is measured before discharge from the delivery room in order to estimate blood loss and to be able to make a comparison with the level of Hb measured in the laboratory as part of clinical routine.
  Interventions: Diagnostic Test: Coagulation tests (TEG, Levels of F1, F2, hs-D-dimer, Plasminogen, PAI 1+2), SpHb before discharge
- vaginal delivery: maternal blood is drawn immediately after the baby's cord is cut and analyzed using thrombelastography with the addition of tranexamic acid. In addition, the following parameters are examined:
  * Levels of Factor 1 (Fibrinogen) and Factor 2 (Thrombin)
  * Level of hs-D-Dimer
  SpHb is measured before discharge from the delivery room in order to estimate blood loss and to be able to make a comparison with the level of Hb measured in the laboratory as part of clinical routine.
  Interventions: Diagnostic Test: Coagulation tests (TEG, Levels of F1, F2, hs-D-dimer, Plasminogen, PAI 1+2), SpHb before discharge

INTERVENTIONS:
Diagnostic Test: Coagulation tests (TEG, Levels of F1, F2, hs-D-dimer, Plasminogen, PAI 1+2), SpHb before discharge — Coagulation tests named earlier as well as SpHb

SUMMARY:
This study aims to find out if there are common major changes in coagulation immediately after delivery of the newborn during Cesarean (C) -section and vaginal birth.

DETAILED DESCRIPTION:
Postpartum Hemorrhage (PPH) is a potentially life-threatening complication of labour and a leading cause of maternal mortality and morbidity. It is defined as a blood loss of 500ml or more in the first 24 hours after birth and it is estimated that about 2% of all parturients are affected. Postpartum hemorrhage is responsible for 8% of maternal deaths in in industrialized nations. The prophylactic use of an uterotonic agent is suggested to reduce the risk of postpartum bleeding.

Tranexamic acid has become another candidate for the prevention of postpartum hemorrhage over the past ten years. It has an antifibrinolytic effect and inhibits hyperfibrinolysis, its clinical effects have been demonstrated in several contexts. In clinical trials outside of obstetrics, tranexamic acid has been found to reduce the need for transfusions during elective procedures and to reduce mortality in patients with extra- or intracranial trauma. In recent studies it is suggested to administer Tranexamic acid already prophylactically during cesarean delivery to reduce blood loss and avoid hyperfibrinolysis and PPH.

What is not known, is how often patients are affected by hyperfibrinolysis during cesarean section and vaginal birth without it manifesting as PPH. In trauma patients, for example, hyperfibrinolysis was found in 5% and moderate hyperfibrinolysis in 57%.

It is unusual to establish a prophylactic treatment without any data on the incidence of the condition, which is aimed to be treated. Therefore, the aim of the study is to provide a data basis for the incidence of hyperfibrinolysis after vaginal delivery and cesarean section.

Primary Aim:

The aim of this study is to quantify the incidence of hyperfibrinolysis during natural birth and C-section. For this purpose, maternal blood is drawn after the baby's cord is cut and analyzed using thrombelastography with the addition of tranexamic acid. In addition, the following parameters are examined:

* Levels of Factor 1 (Fibrinogen) and Factor 2 (Thrombin)
* Level of D-Dimer

Secondary objectives

* Mode of delivery (Vaginal delivery/ C-Section)
* Time cut to delivery as marker for increased manipulation
* Duration of birth in vaginal delivery? Onset of labor until delivery?
* Number of previous births
* Weeks of gestation
* Obstetrical risk factors (multiple gestation, polyhydramnios, prolonged labour, fever)
* Height / weight of parturient
* ASA (American Society of Anesthesiologists) status
* Anticoagulant drugs

At discharge from the delivery room, approximately 6 hours after delivery, hemoglobin levels are checked by noninvasive hemoglobin measurement (Rad-67™ Spot-check Pulse CO-Oximeter® (Masimo Corporation, Irvine, CA) and blood drawing as part of routine clinical practice. In this way, the extent of blood loss can be estimated, and as a further objective the investigators can also verify the usability of spHb (continuous total hemoglobin) measurement in the delivery room.

The usefulness of continuously measuring SpHb in a perioperative setting has previously been described. Several studies have shown that SpHb can help to estimate Hb values in various settings and to reduce unnecessary red blood cell (RBC) transfusions.

In the delivery room setting, the spHb value could serve as an additional tool to reduce unnecessary testing without the cost of overlooking anemic patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older with a singleton or multiple pregnancy who volunteer for the present study and give one blood sample of 6ml

Exclusion Criteria:

1. Age < 18 years
2. Emergency cesarean section
3. History of thrombocytopathy or coagulation disorders
4. Therapy with drugs that influence thrombocyte function and coagulation (ASS less than 5 days ago, clopidogrel, prasugrel, ticagrelor or similar)
5. Lack of consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 780 women after giving birth to a child, 390 in each group
Sampling Method: Non-Probability Sample
Enrollment: 780 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-04-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of Hyperfibrinolysis | immediate after birth
  Ly30-Index is used as marker for Hyperfibrinolysis
D-dimer | immediate after birth
  D-dimer level

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zoidl P, Honnef G, Eichinger M, Eichlseder M, Heuschneider L, Hammer S, Schreiber N, Pruller F, Weiss EC, Amtmann B, Bornemann-Cimenti H. Hyperfibrinolysis During Caesarean Section and Vaginal Delivery: A Prospective Cross-Sectional Study in the Delivery Room. J Clin Med. 2025 Dec 20;15(1):27. doi: 10.3390/jcm15010027. PMID 41517278